CLINICAL TRIAL: NCT01320917
Title: Levonorgestrel-releasing Intrauterine Device Effects on Hemostatic and Arterial Function of Obese Women
Brief Title: Levonorgestrel-releasing Intrauterine Device on Obese Women: Effects on Hemostatic and Arterial Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Rui Alberto Ferriani, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIR-01
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2009-07

CONDITIONS: Contraception Desired; Obesity
Keywords: obesity; contraceptives hormonal; levonorgestrel-releasing intrauterine device; cardiovascular risk
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LNG-IUS (Active Comparator): Insertion of a LNG-IUS device
  Interventions: Device: Levonorgestrel releasing device
- Cu-IUD (Placebo Comparator): Insertion of a Cu-IUD
  Interventions: Device: Cu-IUD insertion

INTERVENTIONS:
Device: Levonorgestrel releasing device — LNG-IUD device releases levonorgestrel in circulation
  Arms: LNG-IUS
Device: Cu-IUD insertion — The action of a Cu-IUD does not release any hormonal compound
  Arms: Cu-IUD

SUMMARY:
Obesity is a disorder associated with metabolic dysfunction and changes in cardiovascular risk markers; the use of oral contraceptives (OCs) may exert a further negative effect on these alterations in patients with PCOS.

To assess the effects on arterial function and structure and hemostatic parameters using an levonorgestrel intrauterine device (IUS-LNG) in women with obesity

A randomized controlled clinical trial.

DETAILED DESCRIPTION:
Setting: Academic hospital.

88 women between 18 and 40 years of age with obesity (BMI between 20 and 40 kg/m2)randomized to use IUS-LNG or Copper-IUD for 12 months

Exclusion criteria: category 3 and 4 Medical Eligibility Criteria for IUD-Cu and IUS-LNG - WHO-2010, pregnancy, lactation, concomitant drugs, smoking.

Main Outcome Measures: Brachial artery flow-mediated vasodilation, carotid intima-media thickness and the carotid artery stiffness index were evaluated at baseline and after 6 and 12 months. Serum markers of cardiovascular disease and hemostatic parameters will be also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 40 years of age with obesity grade I and II who wished to use a contraceptive

Exclusion Criteria:

* any clinical conditions corresponding to category 3 or 4 of the World Health Organization medical eligibility criteria for IUD-LNG or IUD-CU use smoking
* alcoholism
* illicit drug use
* any systemic disease (systemic arterial hypertension, DM, immune system diseases or thyroid diseases) except PCOS
* current or previous (up to two months before the study) use of oral, vaginal, monthly injectable or transdermal combined hormonal contraceptives current or previous use (up to six months before the study) of a long-lasting hormonal contraceptive method (injectable, implant or intrauterine device)
* twelve weeks or less since childbirth
* currently breastfeeding or had stopped breastfeeding within two months of the screening visit
* chronic and/or acute inflammatory processes
* use of drugs known to interfere with inflammatory markers or with CVD risk (anti-androgens, hypoglycemic drugs, anti-inflammatory drugs or statins)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-07 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Arterial function and structure | 6 and 12 months of following
  Brachial artery flow-mediated vasodilation, carotid intima-media thickness and the carotid artery stiffness index

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clinicas de Ribeirao Preto, Departamento Ginecologia e Obstetricia, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Zueff LFN, Melo AS, Vieira CS, Martins WP, Ferriani RA. Cardiovascular risk markers among obese women using the levonorgestrel-releasing intrauterine system: A randomised controlled trial. Obes Res Clin Pract. 2017 Nov-Dec;11(6):687-693. doi: 10.1016/j.orcp.2017.06.001. Epub 2017 Jul 8. PMID 28693985